CLINICAL TRIAL: NCT02717013
Title: The Effect of HMB Supplementation on Adipose Tissue Inflammation and Metabolism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment of subjects.
Sponsor: Metabolic Technologies Inc. (Industry)
Collaborators: Iowa State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: MTI2016-CS01
Record Dates: First submitted 2016-03-11; First posted 2016-03-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Obesity
Keywords: Muscle; Bone; Fat
MeSH Terms: conditions — Obesity; Platelet Glycoprotein IV Deficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo Diet Restriction (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Placebo No Diet Restriction (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- HMB Diet Restriction (Active Comparator)
  Interventions: Dietary Supplement: HMB
- HMB No Diet Restriction (Active Comparator)
  Interventions: Dietary Supplement: HMB

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo capsules containing calcium lactate similar to the HMB capsules.
  Arms: Placebo Diet Restriction; Placebo No Diet Restriction
Dietary Supplement: HMB — HMB capsules supplying 3 grams per day of calcium beta-hydroxyl-beta-methylbutyrate.
  Arms: HMB Diet Restriction; HMB No Diet Restriction

SUMMARY:
This study will determine the effects of supplementing beta-hydroxy-beta-methylbutyrate (HMB) on body composition and strength changes during weight loss. When overweight and obese persons lose weight, and in particular in conjunction with dietary restrictions, muscle, bone mass, and muscle strength are also lost. HMB has been shown to preserve muscle mass and strength, and it is thought that HMB may also preserve muscle, bone, and strength during weight-loss.

DETAILED DESCRIPTION:
Forty obese men (BMI 35-40 kg/m2,18-40 years of age) will be randomly assigned to one of four treatment interventions: 1) Calorie restricted; 2) Calorie restricted and HMB supplemented; 3) No calorie restriction; and 4) No calorie restriction and HMB-supplemented. Over the 8 week interventional period the calorie restricted group is expected to lose 3-5% of initial body weight. Anthropometric measures will be taken weekly, and dual energy x-ray absorptiometry (DXA) body composition and strength will be measured before and after 8-weeks of intervention. Blood and urine will be collected and analyzed at 0, 4, and 8 weeks. Additionally Dietary records and questionnaires concerning quality of life will be administered, and activity will be assessed using questionnaires and pedometers. Muscle biopsies will be taken before and after the 8-week study.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Non-smoker
* Body mass index of 35-40 kg/m2
* Age 18-40 years
* Weight stable for past 6 months (<5 lb. change)
* In good health, free of chronic diseases/conditions that may impact measured outcomes
* Willing and able to consume a weight loss diet
* Willing and able to consume a daily nutritional supplement (in pill form)
* Available for scheduled study commitments during the 2 months of study

Exclusion Criteria:

* Smoke
* Take any cholesterol lowering or weight loss drugs or an drugs or supplements that affect blood lipids, insulin or body composition
* Weigh greater 300 pounds due to weight, size and depth limitations of equipment
* Take dietary supplements
* Have a chronic disease such as:
* Cardiopulmonary disease (e.g. recent myocardial infarction, unstable angina, stroke) or unstable disease
* Severe orthopedic/musculoskeletal or neuromuscular impairments that would contradict exercise
* Sensory impairments that interfere with following directions
* Diagnosis if dementia
* History of malignancy during the past 5 years
* Diabetes mellitus

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Maintenance of bone mineral density | 8 weeks
  Bone mineral density measured by DXA (T-score)
Maintenance of lean mass | 8 weeks
  Lean Mass measured by DXA (kg)
Maintenance of muscle strength | 8 weeks
  Muscle strength will be assessed using a Biodex Isokinetic Dynamometer (N-m)
Maintenance of hand muscle strength | 8 weeks
  Hand muscle strength will be assessed using hand grips (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Valentine, PhD, Principal Investigator — Iowa State University; John A Rathmacher, PhD, Principal Investigator — Metabolic Technologies Inc.
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
No Individual Data will be shared. Data summaries will be available after publication..